CLINICAL TRIAL: NCT00572494
Title: Bioabsorbable Metal Stent Investigation in Chronic Limb Ischemia Treatment
Brief Title: AMS INSIGHT 1 Study - Bioabsorbable Metal Stent Investigation in Chronic Limb Ischemia Treatment
Acronym: AMS-INSIGHT1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Marc Bosiers, MD, AZ Sint-Blasius hospital, Dendermonde, Belgium
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIOTRONIK Reference 27-1
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-02

CONDITIONS: Peripheral Artery Disease
Keywords: Tibial arteries; Absorbable implants; Stents; Limb salvage
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Stenting with AMS
  Interventions: Device: MAGIC EXPLORER (Biotronik AG)
- 2 (Active Comparator): PTA alone
  Interventions: Device: PLEON EXPLORER (Biotronik AG)

INTERVENTIONS:
Device: MAGIC EXPLORER (Biotronik AG) — The lesion is pre-dilated with the PLEON EXPLORER balloon with a length of 10 mm or 15 mm or 20 mm under angiographic control. After dilation, the stenosed area is treated by one AMS implant. If the implanted stent is not fully apposed to the vessel wall or if initial angiography reveals a residual stenosis, the stent may be post-dilated with the delivery system balloon. If necessary, a high-pressure, non-compliant balloon catheter may be used.
  Arms: 1
Device: PLEON EXPLORER (Biotronik AG) — The lesion is dilated with the PLEON EXPLORER balloon with lengths of 10 mm or 15 mm or 20 mm, respectively. In case that the PTA procedure results in a residual stenosis of >50%, the AMS implant should be used to improve the result. A flow-limiting dissection does not qualify for stenting. Best effort must be made to obtain a satisfactory result (e.g. multiple and prolonged inflations) before a patient in the PTA group can be treated with a stent.
  Arms: 2

SUMMARY:
Prospective, multicenter, randomized clinical trial, Follow-up at 1-, 6- and 12 months

This clinical investigation is first of all designed to demonstrate the safety and effectiveness of the MAGIC EXPLORER stent system. The primary objectives of the study are to evaluate the safety and 6-month patency of the bioabsorbable MAGIC EXPLORER stent in patients with stenotic or occlusive atherosclerotic disease of the infrapopliteal arteries. Secondary endpoints are the procedural success, patency at all follow-ups, late lumen loss and limb-salvage rate. Peri-procedural complications (within 24 hours) will be evaluated. Furthermore, data of the balloon catheter PLEON EXPLORER will be collected to demonstrate its effectiveness and safety.

ELIGIBILITY:
Inclusion Criteria:

* Stenotic (> 50%) or occlusive atherosclerotic disease of the infrapopliteal arteries
* Length of lesion < 20mm (less than one stent length)
* Reference vessel diameter should be 3.0-3.5 mm
* A maximum of two lesions in one infrapopliteal vessel treated within the study, or in two vessels of two different legs. (PTA treatment of other infrapopliteal lesions in non-study vessels is allowed outside the study).
* Symptomatic critical limb ischemia (Rutherford 4, 5)
* The patient must be ≥ 50 years.
* Life-expectancy of more than 6 months
* The subject or legal guardian has been informed of the nature of the study; agrees to its provisions and has signed informed consent
* The patient must be available for the appropriate follow-up times for the duration of the study
* The patient is capable to follow all study requirements.

Exclusion Criteria:

* Patient refusing treatment
* The reference segment diameter is not suitable for available stent design
* Length of lesion requires more than one stent implantation
* Previously implanted stent(s) or PTA at the same lesion site
* Lesion lies within or adjacent to an aneurysm
* Inflow-limiting arterial lesions left untreated
* The patient has a known allergy to heparin, Aspirin or other anticoagulant/antiplatelet therapies or a bleeding diatheses or is unable, or unwilling, to tolerate such therapies.
* The patient takes Phenprocoumon (Marcumar).
* The patient has a history of prior life-threatening contrast media reaction.
* The patient is currently enrolled in another investigational device or drug trial.
* The patient is currently breast-feeding, pregnant or intends to become pregnant.
* The patient is mentally ill or retarded.
* The patient is liable for military or civilian service.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2005-07; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Efficacy : patency of the AMS, defined as the absence of a hemodynamically significant restenosis (> 50%) | 6 month
Safety: Complications at 1 month post-procedure (major amputations or any cause of death) | 1 month

SECONDARY OUTCOMES:
Immediate angiographic procedural success, defined as maximal 30% residual stenosis on visual assessment of the planned treatment area. | procedure
Patency at follow-up visits determined with Color Flow Doppler Ultrasound (CFDU) | 1 & 6 months
Late lumen loss at 6 months. | 6 months
Limb-salvage rate at follow-up visits, defined as lack of major amputation. | 1 & 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — AZ Sint-Blasius, Dendermonde, Belgium; Evelyn Diessel, PhD, Study Director — Biotronik SE & Co. KG
Locations (12):
- Austria (3):
  - Medizinische Universität Graz, Graz
  - A.ö. Landeskrankenhaus Klagenfurt, Klagenfurt
  - Allgem. Krankenhaus Vienna, Vienna
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Imelda Ziekenhuis Bonheiden, Bonheiden
  - AZ St-Blasius, Dendermonde
- Germany (5):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Humaine Kliniken Bad Saarow, Bad Saarow
  - Ev. Krankenhaus Herberge Berlin, Berlin
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Mainz, Mainz
- Sint-Elisabeth Ziekenhuis Tilburg, Tilburg, Netherlands